CLINICAL TRIAL: NCT00932776
Title: Tracheobronchial Secretion Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Other Study IDs: AR HSG 268
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Respiration, Artificial; Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Insufficiency

ARMS (2):
- TBA (Experimental)
  Interventions: Device: TBA care device
- Control (Active Comparator)
  Interventions: Device: Control

INTERVENTIONS:
Device: TBA care device — Tracheal suction maneuvers are performed according to the indications provided by the TBA care device or to clinical parameters whichever occurs first.
  Arms: TBA
Device: Control — In this group suction maneuvers are performed according to clinical indications or on a fixed schedule whichever comes first.
  Arms: Control

SUMMARY:
Patients undergoing intubation and mechanical ventilation require removal of secretion by means of trachoebronchial suctioning. Timing of the procedure is mainly based on clinical parameters. TBA Care® is a new commercially available device designed to generate a signal when secretions are present in the respiratory tract of intubated patients, thus indicating the need for endotracheal suctioning only when necessary and prior to clinical deterioration. In a prospective randomized trial in intubated and mechanically ventilated patients of a general ICU the researchers investigated the efficacy of TBA Care® in detecting the presence of retained secretions compared to the standard indicators.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* presence of an endotracheal tube to provide mechanical ventilation
* expected duration of mechanical ventilation greater than 48 hours.

Exclusion Criteria:

* age < 18 years, pregnancy
* presence of active bronchial bleeding

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- A.O. San Gerardo, Monza, MB, Italy

REFERENCES:
- [Derived] Lucchini A, Zanella A, Bellani G, Gariboldi R, Foti G, Pesenti A, Fumagalli R. Tracheal secretion management in the mechanically ventilated patient: comparison of standard assessment and an acoustic secretion detector. Respir Care. 2011 May;56(5):596-603. doi: 10.4187/respcare.00909. Epub 2011 Jan 27. PMID 21276316